CLINICAL TRIAL: NCT05931926
Title: Feasibility and Validation of the Fluispotter®, a Novel Intravenous System for Serial Blood Sampling
Acronym: FLUISPOTTER
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Ulla Feldt-Rasmussen, Professor, Senior Consultant Ulla Feldt-Rasmussen, Rigshospitalet, Denmark
Other Study IDs: FLUISPOTTER
Record Dates: First submitted 2022-08-26; First posted 2023-07-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-06

CONDITIONS: Adrenal Insufficiency
MeSH Terms: conditions — Adrenal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Biospecimen Retention: Samples Without DNA — hormone measurements
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with adrenal insufficiency: 10 patients with adrenal insufficiency due to pituitary desease will be recruited for this arm.
  Interventions: Device: Fluispotter®
- Healthy controls: 10 healthy controls will be recruited for this arm.
  Interventions: Device: Fluispotter®

INTERVENTIONS:
Device: Fluispotter® — The Fluispotter® has been developed for automated extraction, collection and storage of up to 20 dried venous dried blood spot samples of 3-10 μl over the course of up to 20 hours. The system is attached to the patient through a multilumen microcatheter inserted into a peripheral vein in the arm. The Fluispotter will be inserted in both healthy subjects and patients with adrenal insufficiency.

SUMMARY:
The purpose of this study is to test the Fluispotter® technology: A novel system for collection of serial venous samples, which may overcome some of the problems associated with repeated sampling or 20-hour collection of blood samples using standard procedures. The Fluispotter® is the first fully automated, wearable device for obtaining serial blood samples from humans. It is designed to function without operator intervention. The wearable device and - when in place - painless sampling allow sampling during different situations e.g., during sleep, work, play or exercise - whatever the sampling situation requires, including sampling not possible today using wet samples e.g. during everyday activities. Further, it reduces the number of man-hours needed for serial sampling, and minimizes the risks of sample loss, wrong timing, misidentification and contamination.

The primary purpose of this investigator-initiated study is to assess the feasibility, including benefits and harms, of the Fluispotter®, a novel method for serial blood sampling, versus standard blood sampling. The planned setting is a test of the Fluispotter® is a 20-hour period in healthy adults and in adults with secondary adrenal insufficiency due to pituitary disease.

DETAILED DESCRIPTION:
Background In an every-day endocrine setting the dynamic response of hormones is assessed for the diagnosis and evaluation of several conditions such as adrenal insufficiency, Cushing's disease, acromegaly, and growth hormone insufficiency. These procedures require repeated venous sampling. A novel system for collection of serial samples, the Fluispotter®, may overcome some of these problems associated with repeated sampling or 20-hour collection of blood samples. The Fluispotter® is the first fully automated, wearable device for obtaining serial blood samples from humans. It is designed to function without operator intervention. The wearable device and - when in place - painless sampling allow sampling during different situations e.g., during sleep, work, play or exercise - whatever the sampling situation requires, including sampling not possible today using wet samples e.g. during everyday activities. Further, it reduces the number of man-hours needed for serial sampling, and minimizes the risks of sample loss, wrong timing, misidentification and contamination. The dried blood spot technology used in the Fluispotter® was tested for cortisol by comparing with plasma samples and the interassay accuracy and precision were reported to less than 10% across a range of different haematocrit values.

Aim The primary purpose of this investigator-initiated study is to assess the feasibility, including benefits and harms, of the Fluispotter®, a novel method for serial blood sampling, versus standard blood sampling. The planned setting is a test of the Fluispotter® is a 20-hour period in healthy adults and in adults with secondary adrenal insufficiency due to pituitary disease.

The primary outcome for this study is feasibility. This will be assessed using a standardized questionnaire for both staff and participants including items regarding duration of the insertion procedure, ease of insertion, number of re-insertions during the 20-hour study, number of occlusions. Participants will also be asked about perception of pain during insertion, overall acceptance of insertion, acceptance of catheter during the 20-hour admission, and for an overall preference between the new method and conventional blood sampling. In addition, participants will be contacted one week after admission regarding problems related to catheter insertion such as haematomas, pain, infection.

Secondary outcomes will be to assess the validity of cortisol concentrations measured by Dried Blood Spot technology, i.e. the Fluispotter®, compared to the standard blood sampling technique in a clinical setting. Also, Study 1 will compare diurnal cortisol profiles in healthy adults and patients with secondary adrenal insufficiency as well as assessing if the Fluispotter® performs the planned sampling.

Participants In Study 1 a total of 20 individuals will be included, 10 of whom (5 healthy women and 5 healthy men) will constitute the healthy adults and will be recruited through media advertisements.

Five women and 5 men diagnosed with secondary adrenal insufficiency due to pituitary disease will be recruited as patients.These 10 participants will constitute the patient group

The intervention takes place at the Department of Endocrinology and Metabolism at Rigshospitalet, Copenhagen, Denmark.

Sampling Sampling from the Fluispotter® is automatic and does not require attendance from staff. The Fluispotter® will be programmed for 20 samplings at 11:00 am, 13:00 p.m., 17:00 p.m., 21:00 p.m., 23:00 p.m., 00:50 a.m., 02:00 a.m., 02:50 a.m., 04:00 a.m., 04:30 a.m., 05:00 a.m., 05:30 a.m., 06:00 a.m., 06:15 a.m., 06:30 a.m., 06:45 a.m., 07:00 a.m., 07:15 a.m., 07:30 a.m. and 08:00 a.m. The cassettes containing the dried blood spots will be stored at -80◦C until analysis.

Also, eighteen samples from the venous catheter will be drawn at 11:00 am, 13:00 p.m., 17:00 p.m., 21:00 p.m., 23:00 p.m., 01:00 a.m., 03:00 a.m., 04:00 a.m., 04:30 a.m., 05:00 a.m., 05:30 a.m., 06:00 a.m., 06:15 a.m., 06:30 a.m., 06:45 a.m., 07:00 a.m., 07:15 a.m., 07:30 a.m. and 08:00 a.m.

One week after admission the patients will be scheduled for a post-intervention interview. At this visit the patients' arms will be checked for haematomas and the patients will be asked about possible health problems occurring which have arisen after the admission.

ELIGIBILITY:
Healthy subjects

Inclusion Criteria:

* Not receiving regular medication
* Not receiving oral contraceptives or other oestrogens
* No known endocrine or major medical diseases
* No previous surgery of endocrine glands
* No regular smoking
* Not working nightshifts within the last 14 days before assessment
* Able to understand verbal and written instructions in Danish
* Able and willing to sign informed consent
* A negative pregnancy test one-week prior to admission
* Normal infection-, electrolyte- and coagulation-status assessed by standard blood samples

Patients Inclusion criteria

* Adrenal insufficiency due to pituitary disease
* No previous hormone producing pituitary adenomas
* Not receiving oral contraception or other oestrogens
* Stabil pituitary hormone replacement therapy, including hydrocortisone, for the previous three months
* No cardiac, respiratory or lung disease.
* No other disease that potentially requires additional hydrocortisone supplementation
* No regular smoking
* Not working nightshifts within the last 14 days before assessment
* Able to understand verbal and written instructions in Danish
* Able and willing to sign informed consent
* A negative pregnancy test 1-week prior to admission
* Normal infection-, electrolyte- and coagulations-status assessed by standard blood samples

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with secondary pituitary insufficiency
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility - subjects | Day 2-7
  Subjects' acceptance of device - Assessed by a questionnaire consisting of 11 questions designed for this study

SECONDARY OUTCOMES:
Number of succesfull samples by the Fluispotter | Day 2
  The Fluispotter is designed to collect 20 samples during 20 hours. This outcome will describe have many succesful samples the Fluispotter on average performed.
Feasibility - operator | Day 1
  How did the anesthesiologist inserting the Fluispotter catheter percieve the feasibility of the device - Assessed by a questionnaire (uploaded)

OTHER OUTCOMES:
Increase of cortisol due to sampling stress | through study completion, an average of 1 year
  The samples obtained from the Fluispotter willl be compared with wet samples prior to and after collection of samples. Any difference could be attribued to sampling stress.

CONTACTS AND LOCATIONS:
Overall Officials: Ulla Feldt-Rasmussen, Prof, Principal Investigator — Rigshospitalet, Denmark

IPD SHARING:
Plan to Share IPD: No
There are currently no plan to share IPD with other researchers

REFERENCES:
- [Background] Ollerenshaw JD, Schroder M, Velschow S. A novel device for serial venous blood sampling in a canine model. J Pharmacol Toxicol Methods. 2022 Mar-Apr;114:107155. doi: 10.1016/j.vascn.2022.107155. Epub 2022 Jan 14. PMID 35038558
- [Background] Adhikari KB, Rohde M, Velschow S, Feldt-Rasmussen U, Johannesen J, Johnsen AH. Fluispotter, a novel automated and wearable device for accurate volume serial dried blood spot sampling. Bioanalysis. 2020 May;12(10):665-681. doi: 10.4155/bio-2020-0048. Epub 2020 Jun 3. PMID 32489105